CLINICAL TRIAL: NCT03013179
Title: Intergenerational Impact of Genetic and Psychological Factors on Blood Pressure
Brief Title: Intergenerational Blood Pressure Study
Acronym: InterGEN
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: 1311012986; 5R01NR013520 (NIH)
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sample for DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Black/African American Women and their 3-5 year old children

SUMMARY:
This project, the Intergenerational Blood Pressure Study, is a 5 year research study funded by the National Institutes of Health/National Institute of Nursing Research and led by the Yale University School of Nursing and The Consultation Center at the Yale University School of Medicine, Department of Psychiatry in partnership with Head Start programs across CT. The investigators seek to reduce hypertension health disparities among underserved Black/African American children and their mothers by conducting community-based research to better understand the genetic, psychological, and environmental factors that may contribute to high blood pressure.

DETAILED DESCRIPTION:
This study will examine: (1) the impact of (GXE) genetic and psychological environmental factors (discrimination, depression, and parenting behaviors) on the health of African American (AA) children aged 3 through 5 years and (2) the GXE risk for hypertension (HTN) in AA women and children. The overall goal of this project is to delineate the psychobiological (GXE interaction) mechanisms through which AA mothers' perceived racial discrimination, mental health, and parenting behavior affect their own and their young children's blood pressure (BP) over time. The research will examine both genetic (candidate gene and epigenetic effects) and psychological (maternal perceived racial discrimination, mental health, and parenting behavior) interaction effects on BP on this population. The investigators will employ a psychobiological approach by: utilizing psychological and biological assessments using a longitudinal cohort research design, a 2-step candidate gene and epigenetic methodology, and use of ancestry informative markers to account for population stratification admixture to explore GXE interactions on BP in AA mothers and children. Data analysis for the study will be conducted using multiple mixed modeling, cross-validation, and false discovery rate methods. The investigators will enroll 250 AA children aged 3 through 5 years and their (n=250) mothers/maternal caregivers. The investigators will assess mother and child factors every six months for 2 years. The investigators propose the following: Aim 1: Examine the GXE interaction and epigenetic effects of mothers' perceived racial discrimination and its influence on BP over a period of two years. Aim 2: Examine the GXE interaction and epigenetic effects of mothers' mental health status [symptoms of depression] and its influence on BP over a period of two years. Aim 3: Examine the GXE interaction and epigenetic effects of mothers' parenting behavior and its influence on BP over a period of two years. This project supports the National Institute of Nursing Research mission "to promote and improve the health of individuals, families, communities, and populations" by conducting basic research on the health and illness of women and young children. The proposed research extends nursing science by integrating the biological (genetics) and behavioral (psychology) components that can inform the combination of multi-level factors that contribute to AAs having the highest incidence of HTN in the US. Findings from this project can contribute to developing interventions that address genetic and psychological factors to reduce these risks for HTN.

ELIGIBILITY:
Inclusion Criteria:

Mothers must:

* Self-identify as Black/African American
* Be 21 years or older
* Have a 3-5 year old biological child
* Not be impaired by a though disorder, psychosis, or mania
* Confirm that their child will be able to provide saliva sample for DNA
* Be English-speaking

Exclusion Criteria:

* None

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Black/African American women and their 3-5 year old children in CT
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 18 months
  Manual blood pressure taken according to JNC-7 guidelines, average of 3 resting blood pressure measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Y Taylor, PhD, Principal Investigator — Yale University; Cindy A Crusto, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Nursing, Orange, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Genomic Data Sharing Plan in place, in accordance with NIH regulations Only de-identified genomic data will be shared with dbGaP, to which other researchers will be able to apply for access. Data will be submitted within 1 year after analyses are complete.

REFERENCES:
- [Background] Taylor JY, Wright ML, Crusto CA, Sun YV. The Intergenerational Impact of Genetic and Psychological Factors on Blood Pressure (InterGEN) Study: Design and Methods for Complex DNA Analysis. Biol Res Nurs. 2016 Oct;18(5):521-30. doi: 10.1177/1099800416645399. Epub 2016 Apr 26. PMID 27118148
- [Background] Crusto CA, Barcelona de Mendoza V, Connell CM, Sun YV, Taylor JY. The Intergenerational Impact of Genetic and Psychological Factors on Blood Pressure Study (InterGEN): Design and Methods for Recruitment and Psychological Measures. Nurs Res. 2016 Jul-Aug;65(4):331-8. doi: 10.1097/NNR.0000000000000163. PMID 27362519
- [Background] Barcelona de Mendoza V, Wright ML, Agaba C, Prescott L, Desir A, Crusto CA, Sun YV, Taylor JY. A Systematic Review of DNA Methylation and Preterm Birth in African American Women. Biol Res Nurs. 2017 May;19(3):308-317. doi: 10.1177/1099800416669049. Epub 2016 Sep 19. PMID 27646016
- See also: Click here for more information about this study: Intergenerational Blood Pressure Study — http://intergen.yale.edu/